CLINICAL TRIAL: NCT01298544
Title: A Phase 4, Open-label Study to Evaluate Persistence of the Antibody Response Elicited by Prevenar in Healthy Children in China Who Have Been Previously Immunized With a 4-dose Series of a Pneumococcal Conjugate Vaccine During Infancy in Study 0887x-101518
Brief Title: A Study to Assess the Antibody Response of Healthy Chinese Children Who Have Been Vaccinated Previously With 4-doses of Prevenar (a Pneumococcal Vaccine) as Babies and Toddlers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1841009; 6114A1-4001
Record Dates: First submitted 2010-11-29; First posted 2011-02-17 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Pneumococcal Disease
Keywords: Vaccine; Prevenar; Pneumococcal disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Other)
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — One 5mL blood draw for immunogenicity at least 3 years post completion of clinical study 0887X-101518.

SUMMARY:
In 2005, Wyeth conducted study 0887X-101518 (NCT00488826) in which Chinese infants received either Prevenar alone (Group 1), Prevenar given with a Diphtheria, Tetanus and acellular Pertussis (DTaP) vaccine (Group 2) or DTaP alone (Group 3). This follow up study (at least 3 years after the last vaccination) will assess the antibody concentrations in children who previously completed Wyeth study 0887X-101518.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who participated in and completed Wyeth study 0887X 101518.
* Healthy subject as determined by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

* Vaccination with any licensed or investigational pneumococcal vaccine since completion of Wyeth study 0887X 101518.
* History of culture proven invasive disease caused by S pneumoniae since the completion of Wyeth study 0887X 101518.
* Known or suspected immune deficiency or suppression since participation in Wyeth study 0887X 101518.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 335 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- China (10):
  - Chengxiang Town Hospital, Longan County, Guangxi
  - Longan County CDC, Longan County, Guangxi
  - Nanyu Town Hospital, Longan County, Guangxi
  - Yanjiang Town Hospital, Longan County, Guangxi
  - Natong Town Hospital, Longan County, Guangxi
  - Qiaojian Town Hospital, Longan County, Guangxi
  - Gutan Village Hospital, Longan County, Guangxi
  - Dingdang Town Hospital, Longan County, Guangxi
  - Yangwan Hospital, Longan County, Guangxi
  - GuangXi Center for Disease Prevention and Control, Nanning, Guangxi

REFERENCES:
- [Derived] Li R, Fang KX, Young M Jr, Zhou X, Chen Z, Liang JZ, Giardina PC, Scott DA. Long-term antibody persistence study (3 years after last dose) of the 7-valent pneumococcal conjugate vaccine in young children in China. Vaccine. 2016 Oct 17;34(44):5359-5365. doi: 10.1016/j.vaccine.2016.08.070. Epub 2016 Sep 8. PMID 27616471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible participants who completed a previous study, 0887X-101518 (NCT00488826), were invited to participate in this study, at a timepoint at least 3 years after their last vaccination in study 0887X-101518.
Pre-assignment Details: No vaccines administered during study. However, participants assessed according to the vaccine group they were assigned to in study 0887X-101518: 7-valent pneumococcal conjugate vaccine (7vPnC) alone (Group 1), 7vPnC given concomitantly with diphtheria, tetanus, and acellular pertussis vaccine (DTaP) (Group 2), or DTaP alone (Group 3).
Groups:
- Entire Study Population: All randomized participants
Period: Overall Study
Arm/Group | Entire Study Population
Started | 335
Completed | 335
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.04 (0.150)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 186

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody, 36 Months After the Toddler Dose
Description: Antibody geometric mean concentration (GMC) as measured by mcg/mL for 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F). GMC (7vPnC, 7vPnC/DTaP, and DTap) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: Day 1 (36 months after toddler dose)
Population: Evaluable Immunogenicity population: eligible participants who had blood drawn within required time frame, had at least 1 valid and determinate assay result for the proposed analysis, received no prohibited vaccines, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Groups:
- 7vPnC: No investigational product was administered during the study. Participants previously received 7-valent pneumococcal conjugate vaccine (7vPnC) in a preceding study, 0887X-101518, at 3 months (vaccination 1), 4 months (vaccination 2), 5 months (vaccination 3), and 12 to 15 months (vaccination 4) of age.
- 7vPnC and DTaP: No investigational product was administered during the study. Participants previously received 7vPnC concomitantly with diphtheria, tetanus, and acellular pertussis vaccine (DTaP) in a preceding study, 0887X-101518, at 3 months (vaccination 1), 4 months (vaccination 2), 5 months (vaccination 3), and 12 to 15 months (vaccination 4) of age.
- DTaP Alone: No investigational product was administered during the study. Participants previously received DTaP in a preceding study, 0887X-101518, at 3 months (vaccination 1), 4 months (vaccination 2), and 5 months (vaccination 3).
Arm/Group | 7vPnC | 7vPnC and DTaP | DTaP Alone
Number analyzed (Participants) | 123 | 121 | 91
microgram per milliliter (mcg/mL)
  Serotype 4 | 0.98 [0.77 to 1.23] | 0.66 [0.52 to 0.84] | 0.41 [0.29 to 0.58]
  Serotype 6B | 11.35 [9.71 to 13.27] | 9.24 [7.66 to 11.16] | 3.37 [2.76 to 4.13]
  Serotype 9V | 1.35 [1.13 to 1.62] | 1.29 [1.08 to 1.54] | 1.05 [0.83 to 1.32]
  Serotype 14 | 4.50 [3.38 to 5.98] | 3.02 [2.25 to 4.05] | 0.55 [0.40 to 0.76]
  Serotype 18C | 0.80 [0.66 to 0.97] | 0.77 [0.60 to 0.98] | 0.34 [0.24 to 0.47]
  Serotype 19F | 10.14 [8.06 to 12.75] | 5.67 [4.50 to 7.14] | 1.70 [1.35 to 2.15]
  Serotype 23F | 3.31 [2.80 to 3.91] | 2.71 [2.26 to 3.25] | 1.44 [1.17 to 1.76]
Statistical Analysis 1: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 4; Test type: Superiority or Other; Ratio of GMCs = 0.68, 95% CI 2-sided [0.48 to 0.94] — Calculated by back transforming the ratio difference between vaccine groups on logarithmic scale. Back transformations of CIs based on Student t distribution for ratio difference of the logarithms of the measures (Group 2-Group 1)
Statistical Analysis 2: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 6B; Test type: Superiority or Other; Ratio of GMCs = 0.81, 95% CI 2-sided [0.64 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 9V; Test type: Superiority or Other; Ratio of GMCs = 0.95, 95% CI 2-sided [0.74 to 1.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 14; Test type: Superiority or Other; Ratio of GMCs = 0.67, 95% CI 2-sided [0.45 to 1.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 18C; Test type: Superiority or Other; Ratio of GMCs = 0.96, 95% CI 2-sided [0.70 to 1.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 19F; Test type: Superiority or Other; Ratio of GMCs = 0.56, 95% CI 2-sided [0.40 to 0.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 23F; Test type: Superiority or Other; Ratio of GMCs = 0.82, 95% CI 2-sided [0.64 to 1.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 4; Test type: Superiority or Other; Ratio of GMCs = 1.97, 95% CI 2-sided [1.39 to 2.80] — Calculated by back transforming the ratio difference between vaccine groups on logarithmic scale. Back transformations of CIs based on Student t distribution for ratio difference of the logarithms of the measures (Groups 1 and 2 combined-Group 3)
Statistical Analysis 9: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 6B; Test type: Superiority or Other; Ratio of GMCs = 3.04, 95% CI 2-sided [2.41 to 3.84] — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 10: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 9V; Test type: Superiority or Other; Ratio of GMCs = 1.26, 95% CI 2-sided [0.98 to 1.62] — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 11: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 14; Test type: Superiority or Other; Ratio of GMCs = 6.66, 95% CI 2-sided [4.53 to 9.79] — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 12: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 18C; Test type: Superiority or Other; Ratio of GMCs = 2.34, 95% CI 2-sided [1.68 to 3.24] — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 13: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 19F; Test type: Superiority or Other; Ratio of GMCs = 4.47, 95% CI 2-sided [3.29 to 6.07] — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 14: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 23F; Test type: Superiority or Other; Ratio of GMCs = 2.08, 95% CI 2-sided [1.65 to 2.63] — [estimate comment as in outcome 1, analysis 8]

2. Other Pre Specified Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 mcg/mL, 36 Months After the Toddler Dose
Description: Percentage of participants achieving predefined antibody threshold ≥0.35 mcg/mL along with the corresponding 95% CI for the 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F). Exact 2-sided CI based on the observed proportion of participants.
Time Frame: Day 1 (36 months after toddler dose)
Population: Evaluable Immunogenicity population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 7vPnC | 7vPnC and DTaP | DTaP Alone
Number analyzed (Participants) | 123 | 121 | 91
Percentage of participants
  Serotype 4 | 82.9 [75.1 to 89.1] | 64.5 [55.2 to 73.0] | 48.8 [37.7 to 60.0]
  Serotype 6B | 100.0 [97.0 to 100.0] | 100.0 [97.0 to 100.0] | 97.8 [92.3 to 99.7]
  Serotype 9V | 93.5 [87.6 to 97.2] | 94.2 [88.4 to 97.6] | 83.5 [74.3 to 90.5]
  Serotype 14 | 95.1 [89.7 to 98.2] | 91.7 [85.3 to 96.0] | 63.7 [53.0 to 73.6]
  Serotype 18C | 81.3 [73.3 to 87.8] | 69.4 [60.4 to 77.5] | 45.5 [34.8 to 56.4]
  Serotype 19F | 100.0 [97.0 to 100.0] | 97.5 [92.9 to 99.5] | 92.2 [84.6 to 96.8]
  Serotype 23F | 100.0 [97.0 to 100.0] | 99.2 [95.5 to 100.0] | 93.4 [86.2 to 97.5]
Statistical Analysis 1: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 4; Test type: Superiority or Other; Difference in proportions = -18.5, 95% CI 2-sided [-29.4 to -7.3] — Difference in proportions, expressed as a percentage. Exact 2 sided CI for the difference in proportions (Group 2-Group 1), expressed as a percentage
Statistical Analysis 2: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 6B; Test type: Superiority or Other; Difference in proportions = 0.0, 95% CI 2-sided [-3.1 to 3.0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 9V; Test type: Superiority or Other; Difference in proportions = 0.7, 95% CI 2-sided [-5.9 to 7.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 14; Test type: Superiority or Other; Difference in proportions = -3.4, 95% CI 2-sided [-10.3 to 3.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 18C; Test type: Superiority or Other; Difference in proportions = -11.9, 95% CI 2-sided [-22.7 to -1.0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 19F; Test type: Superiority or Other; Difference in proportions = -2.5, 95% CI 2-sided [-7.1 to 0.6] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 7vPnC vs 7vPnC and DTaP; Serotype 23F; Test type: Superiority or Other; Difference in proportions = -0.8, 95% CI 2-sided [-4.5 to 2.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 4; Test type: Superiority or Other; Difference in proportions = 25.0, 95% CI 2-sided [12.7 to 37.0] — Difference in proportions, expressed as a percentage. Exact 2 sided CI for the difference in proportions (Group 1 and 2 combined-Group 3), expressed as a percentage
Statistical Analysis 9: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 6B; Test type: Superiority or Other; Difference in proportions = 2.2, 95% CI 2-sided [-0.011 to 7.715] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 10: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 9V; Test type: Superiority or Other; Difference in proportions = 10.3, 95% CI 2-sided [1.9 to 19.6] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 11: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 14; Test type: Superiority or Other; Difference in proportions = 29.7, 95% CI 2-sided [19.4 to 40.5] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 12: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 18C; Test type: Superiority or Other; Difference in proportions = 30.0, 95% CI 2-sided [17.9 to 41.5] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 13: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 19F; Test type: Superiority or Other; Difference in proportions = 6.5, 95% CI 2-sided [1.2 to 13.9] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 14: Comparison: 7vPnC vs 7vPnC and DTaP vs DTaP Alone; Serotype 23F; Test type: Superiority or Other; Difference in proportions = 6.2, 95% CI 2-sided [1.8 to 13.0] — [estimate comment as in outcome 2, analysis 8]

ADVERSE EVENTS:
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/335
Other Adverse Events (participants affected / at risk) | 0/335

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.